CLINICAL TRIAL: NCT04528225
Title: Hypothyroidism After Postoperative Radiation Therapy in Patients With Breast Cancer：a Prospective Clinical Study
Brief Title: A Prospective Study of Hypothyroidism After Radiotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, professor of medicine, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC2444
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2020-08

CONDITIONS: Breast Neoplasms; Hypothyroidism; Radiation Toxicity
MeSH Terms: conditions — Breast Neoplasms; Hypothyroidism; Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to prospectively investigate the incidence of hypothyroidism after postoperative radiotherapy and identify risk factors for development of hypothyroidism. Patients with breast cancer treated with surgery followed by radiotherapy is enrolled. Thyroid function was assessed at baseline and different times after radiotherapy. The radiation technique, thyroid dose parameters and hypothyroidism are prospective evaluated, and the dose-effect relationship is analyzed.

DETAILED DESCRIPTION:
Breast cancer patients treated with radiotherapy after surgery are prospectively enrolled. Thyroid function is evaluated mainly by the measurement of thyroid-stimulating hormone (TSH), free triiodo-thyronine (FT3) and free thyroxine (FT4). Thyroid function is regularly assessed before and after radiotherapy. The radiation technique and thyroid dose parameters are assessed. Development of subclinical or biochemical hypothyroidism is noted. The incidence and risk factors of hypothyroidism is analyzed. The dose-volume constraints that correlate with functional impairment of the thyroid in breast cancer patients treated with radiotherapy is discussed.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer patients at first diagnosis, patients who are treated with radiotherapy after breast conserving surgery or modified radical mastectomy, no medical history of hyperthyroidism, hypothyroidism or thyroiditis, have never taken thyroxine, no thyroid surgery.

Exclusion Criteria:

Absence or ectopic thyroid gland, previous radiotherapy of the neck, diseases of thalamus or pituitary, previous radiotherapy of thalamus or pituitary

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients treated with radiotherapy after surgery are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related hypothyroidism as assessed by CTCAE v4.0 | up to 2 years
  The subclinical and biochemical hypothyroidism are regularly assessed with the measurement of thyroid-stimulating hormone (TSH), free triiodo-thyronine (FT3) and free thyroxine (FT4).

CONTACTS AND LOCATIONS:
Overall Officials: Shu-lian Wang, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China